CLINICAL TRIAL: NCT00398879
Title: A Randomized Placebo-Controlled Study of Perifosine in Combination With Single Agent Chemotherapy for Metastatic Cancer Patients
Brief Title: Placebo-Controlled Study of Perifosine + Single Agent Chemotherapy for Metastatic Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Perifosine 211
Record Dates: First submitted 2006-11-06; First posted 2006-11-14 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2012-02

CONDITIONS: Colon Cancer
Keywords: Capecitabine
MeSH Terms: conditions — Colonic Neoplasms | interventions — perifosine; Capecitabine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Perifosine + Capecitabine (Experimental): Perifosine 50 mg/d qd + Capecitabine 825 mg/m^2 BID days 1 - 14 q 3 weeks until progression
  Interventions: Drug: Perifosine; Drug: Capecitabine
- Arm 2: Perifosine Placebo + Capecitabine (Placebo Comparator): Perifosine Placebo 50 mg/d qd + Capecitabine 825 mg/m^2 BID days 1 - 14 q 3 weeks until progression
  Interventions: Drug: Capecitabine; Other: Perifosine Placebo

INTERVENTIONS:
Drug: Perifosine — Perifosine 50 mg/d qd
  Other Names: D-21266; KRX-0401
  Arms: Arm 1: Perifosine + Capecitabine
Drug: Capecitabine — Capecitabine 825 mg/m^2 BID days 1 - 14 q 3 weeks
Other: Perifosine Placebo — Placebo to Perifosine 50 mg/d qd
  Other Names: placebo
  Arms: Arm 2: Perifosine Placebo + Capecitabine

SUMMARY:
This is an exploratory phase 2, randomized placebo-controlled trial with stratification for disease and chemotherapy type. The study is subsequently closed to enrollment in all arms except patients with metastatic colorectal cancer which would be randomized to either capecitabine plus perifosine or capecitabine alone.

The effects of perifosine may be manifested by increased time to progression, tumor regression reflected in partial or complete responses, or a combination of these outcomes. The primary goal of this trial is to obtain a preliminary and objective assessment of the effects of perifosine on time to progression.

DETAILED DESCRIPTION:
This is an exploratory phase 2, randomized placebo-controlled trial with stratification for disease and chemotherapy type. If there is any evidence of improved time to progression in any tumor type with any of the drugs to be evaluated, the initial study or component(s) of the study will be expanded to increase the certainty that this is an effect of perifosine. If there is compelling evidence of benefit from this study, a phase 3 trial will be conducted to obtain proof of principle.

Primary Study Objectives:

To determine the time to tumor progression when receiving single agent chemotherapy (capecitabine) in combination with perifosine in comparison to patients receiving single agent chemotherapy (capecitabine) alone (i.e., with placebo).

Secondary Study Objectives:

* To determine the toxicity of single agent chemotherapy in combination with perifosine.
* To compare the time to progression of chemotherapy in combination with placebo to historical experience.
* Overall survival will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the treating physician, treatment with one of the following regimens should represent an appropriate treatment for the patient.

   - Capecitabine 825 mg/m2 BID days 1 - 14 q 3 weeks
2. Patients should have a histologically or cytologically confirmed diagnosis of colorectal cancer.
3. Patients must have received at least one but no more than two prior chemotherapy regimen(s) for the treatment of metastatic or recurrent disease.
4. ECOG performance status 0 or 1.

   * Leukocytes >= 4,000/μL
   * absolute neutrophil count >= 1,500/ μL
   * platelets >= 100,000/ μL
   * HCT > 28% (with or without growth factor support)
   * Creatinine <= 2.5 mg/dl
   * total bilirubin < 1.5 x upper limit of normal
   * transaminase < 2.5 x upper limit of normal
5. Patients must have recovered from acute toxicity-excluding alopecia-related to prior therapy, including surgery or radiotherapy.
6. Patients with brain metastases may be admitted, provided the disease has been treated and been stable for 2 months.
7. Patients must have ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients receiving any other investigational agents or devices.
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to perifosine (miltefosine or edelfosine).
3. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, psychiatric illness, or social situations that would limit compliance with study requirements.
4. HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study due to potential pharmacokinetic interactions with perifosine.
5. Patients with a history of unstable or newly diagnosed angina pectoris, recent myocardial infarction (within 6 months of enrollment), or New York Heart Assoc. class II - IV congestive heart failure.
6. Female patients who are pregnant or lactating are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2005-08; Primary Completion 2010-12 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Effects of perifosine on time to progression | Every 12 weeks
  Time to progression will be measured from the first day of study drug until progression.

SECONDARY OUTCOMES:
Toxicity | Every 12 weeks
  Determination of the toxicity of single agent chemotherapy in combination with perifosine. Toxicity evaluation is to be performed throughout the study.
Comparison of time to progression to historical experience | Every 12 weeks
  To compare the time to progression of chemotherapy in combination with placebo to historical experience.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Henderson, MD, Study Chair — Online Collaborative Oncology Group
Locations (48):
- United States (48):
  - AOI Pharmaceuticals Investigative Site, Tucson, Arizona
  - AOI Pharmaceuticals Investigative Site, Beverly Hills, California
  - AOI Pharmaceuticals Investigative Site, Deer Park, California
  - AOI Pharmaceuticals Investigative Site, Monterey, California
  - AOI Pharmaceuticals Investigative Site, Newport Beach, California
  - AOI Pharmaceuticals Investigative Site, Pomona, California
  - AOI Pharmaceuticals Investigative Site, Santa Rosa, California
  - AOI Pharmaceuticals Investigative Site, Soquel, California
  - AOI Pharmaceuticals Investigative Site, Stockton, California
  - AOI Pharmaceuticals Investigative Site, Colorado Springs, Colorado
  - AOI Pharmaceuticals Investigative Site, Greeley, Colorado
  - AOI Pharmaceuticals Investigative Site, Middletown, Connecticut
  - AOI Pharmaceuticals Investigative Site, Norwich, Connecticut
  - AOI Pharmaceuticals Investigative Site, Aventura, Florida
  - AOI Pharmaceuticals Investigative Site, Coral Springs, Florida
  - AOI Pharmaceuticals Investigative Site, Lake City, Florida
  - AOI Pharmaceuticals Investigative Site, Miami, Florida
  - AOI Pharmaceuticals Investigative Site, Ormond Beach, Florida
  - AOI Pharmaceuticals Investigative Site, Sebastian, Florida
  - AOI Pharmaceuticals Investigative Site, Vero Beach, Florida
  - AOI Pharmaceuticals Investigative Site, Augusta, Georgia
  - AOI Pharmaceuticals Investigative Site, Lawrenceville, Georgia
  - AOI Pharmaceuticals Investigative Site, Marietta, Georgia
  - AOI Pharmaceuticals Investigative Site, Galesburg, Illinois
  - AOI Pharmaceuticals Investigative Site, Park Ridge, Illinois
  - AOI Pharmaceuticals Investigative Site, Louisville, Kentucky
  - AOI Pharmaceuticals Investigative Site, Lafayette, Louisiana
  - AOI Pharmaceuticals Investigative Site, Grand Rapids, Michigan
  - AOI Pharmaceuticals Investigative Site, Kalamazoo, Michigan
  - AOI Pharmaceuticals Investigative Site, Branson, Missouri
  - AOI Pharmaceuticals Investigative Site, Billings, Montana
  - AOI Pharmaceuticals Investigative Site, Great Falls, Montana
  - AOI Pharmaceuticals Investigative Site, Albany, New York
  - AOI Pharmaceuticals Investigative Site, Armonk, New York
  - AOI Pharmaceuticals Investigative Site, Great Neck, New York
  - AOI Pharmaceuticals Investigative Site, Wilmington, North Carolina
  - AOI Pharmaceuticals Investigative Site, Dayton, Ohio
  - AOI Pharmaceuticals Investigative Site, Pottsville, Pennsylvania
  - AOI Pharmaceuticals Investigative Site, Sayre, Pennsylvania
  - AOI Pharmaceuticals Investigative Site, Greenville, South Carolina
  - AOI Pharmaceuticals Investigative Site, Chattanooga, Tennessee
  - AOI Pharmaceuticals Investigative Site, Memphis, Tennessee
  - AOI Pharmaceuticals Investigative Site, Dallas, Texas
  - AOI Pharmaceuticals Investigative Site, Tyler, Texas
  - AOI Pharmaceuticals Investigative Site, Chesapeake, Virginia
  - AOI Pharmaceuticals Investigative Site, Norfolk, Virginia
  - AOI Pharmaceuticals Investigative Site, Spokane, Washington
  - AOI Pharmaceuticals Investigative Site, Appleton, Wisconsin

REFERENCES:
- [Result] Bendell JC, Nemunaitis J, Vukelja SJ, Hagenstad C, Campos LT, Hermann RC, Sportelli P, Gardner L, Richards DA. Randomized placebo-controlled phase II trial of perifosine plus capecitabine as second- or third-line therapy in patients with metastatic colorectal cancer. J Clin Oncol. 2011 Nov 20;29(33):4394-400. doi: 10.1200/JCO.2011.36.1980. Epub 2011 Oct 3. PMID 21969495